CLINICAL TRIAL: NCT04294836
Title: Randomized Phase II Clinical Trial of Oral Turmeric Supplementation in Patients With Advanced Cervical Cancer
Brief Title: Curcumin in Advanced Cervical Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Issues with local regulatory authority
Sponsor: Instituto Nacional de Cancerologia, Columbia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IX-023435
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2020-06

CONDITIONS: Cervical Cancer, Stage IIB
Keywords: curcumin; natural antioxidant
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Phase II clinical trial, randomized and placebo controlled
Who Masked: Participant, Investigator
Masking Description: double blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curcumin (Experimental): Chemotherapy (cisplatin) plus concomitant radiation therapy (teletherapy + high or low rate brachytherapy) + Curcugreen (BCM95) 2000mg daily (each 6h)
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator): Chemotherapy (cisplatin) plus concomitant radiation therapy (teletherapy + high or low rate brachytherapy) + Placebo Capsules 500mg 2000mg daily (each 6h)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Curcumin — BCM-95® (CURCUGREEN®) is a 100 percent pure extract of turmeric with enhanced bio-availability and bio-efficacy. Its powerful health-promoting benefits are derived from the colorful and aromatic qualities of the Indian spice
  Arms: Curcumin
Drug: Placebo oral tablet — PLACEBO Capsules 500mg
  Arms: Placebo

SUMMARY:
Determine the efficacy and safety of turmeric in the treatment of patients with advanced cervical cancer. Efficacy will be determined through radiological and histopathological criteria through the rate of response to treatment, duration of response, the rate of objective response and disease control, as well as overall survival and disease-free survival. The safety of therapy will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) classification

DETAILED DESCRIPTION:
A placebo-controlled phase II clinical trial will be developed in patients with advanced cervical cancer who have an indication for radiotherapy. Those who accept to participate will receive the standard treatment with established chemo-radiation and will be randomized in two arms, the experimental will receive 500mg of the commercial presentation (curcugreen) c / 6h VO x 16 weeks and the control arm will receive placebo. The operative hypotheses are: the addition of curcumin to the treatment improves the cumulative probability of 3-year overall survival by 20% and improves the treatment response rate. The statistical analysis will include a Cox proportional hazards model and the results of the groups will be compared with the Student's T-test or ANOVA. This research hopes to collect tissue samples for future research that allows the identification of predictive biomarkers and disease prognoses.

ELIGIBILITY:
Inclusion Criteria:

Women aged 18 years or older

* Voluntary acceptance of participation and signing of informed consent
* Radiotherapy indication
* Histological confirmation of squamous cervical cancer or histologically confirmed adenocarcinoma
* Stage IIB - VAT
* Chemo-radiation indication with Cisplatin, Cisplatin/fluorouracil, Carboplatin (if cisplatin intolerant)
* ECOG equal to or less than 1 and a Karnofsky index equal to or greater than 70%.

Exclusion Criteria:

* Being pregnant or breastfeeding
* Presence of second concomitant neoplasia
* Any previous surgical, radiotherapy or chemotherapy treatment.
* Diagnosis of invasive recurrent carcinoma of the cervix
* Receive anticoagulant therapy
* Receive immunosuppression therapy
* Presence of coagulation disorders, such as platelet count less than 100,000 at the time of the joint evaluation, absolute neutrophil count less than 1,500 / ml
* Presence of signs of systemic infection
* Renal failure, creatinine clearance less than 45 ml/min confirmed with glomerular filtration less than 45 ml / min; evidence of unilateral renal exclusion
* Patients with uncontrolled metabolic disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare overall survival and progression free survival | 3 yr
  Global survival
Compare the objective response rate using RECIST radiological criteria | 1 yr
  Objective response by RECIST criteria
Compare the disease control rate | 1 yr
  Disease control rate

SECONDARY OUTCOMES:
Describe the safety of research therapy by classifying Common Terminology Criteria for Adverse Events (CTCAE) | 1 yr
  Common Terminology Criteria for Adverse Events (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Carreño, Md, Principal Investigator — Instituto Nacional de Cancerologia de Mexico

REFERENCES:
- [Result] Saadipoor A, Razzaghdoust A, Simforoosh N, Mahdavi A, Bakhshandeh M, Moghadam M, Abdollahi H, Mofid B. Randomized, double-blind, placebo-controlled phase II trial of nanocurcumin in prostate cancer patients undergoing radiotherapy. Phytother Res. 2019 Feb;33(2):370-378. doi: 10.1002/ptr.6230. Epub 2018 Nov 14. PMID 30427093
- [Result] Javvadi P, Segan AT, Tuttle SW, Koumenis C. The chemopreventive agent curcumin is a potent radiosensitizer of human cervical tumor cells via increased reactive oxygen species production and overactivation of the mitogen-activated protein kinase pathway. Mol Pharmacol. 2008 May;73(5):1491-501. doi: 10.1124/mol.107.043554. Epub 2008 Feb 5. PMID 18252805
- [Result] Javvadi P, Hertan L, Kosoff R, Datta T, Kolev J, Mick R, Tuttle SW, Koumenis C. Thioredoxin reductase-1 mediates curcumin-induced radiosensitization of squamous carcinoma cells. Cancer Res. 2010 Mar 1;70(5):1941-50. doi: 10.1158/0008-5472.CAN-09-3025. Epub 2010 Feb 16. PMID 20160040
- [Result] Hejazi J, Rastmanesh R, Taleban FA, Molana SH, Hejazi E, Ehtejab G, Hara N. Effect of Curcumin Supplementation During Radiotherapy on Oxidative Status of Patients with Prostate Cancer: A Double Blinded, Randomized, Placebo-Controlled Study. Nutr Cancer. 2016;68(1):77-85. doi: 10.1080/01635581.2016.1115527. Epub 2016 Jan 15. PMID 26771294
- [Result] Sasaki H, Sunagawa Y, Takahashi K, Imaizumi A, Fukuda H, Hashimoto T, Wada H, Katanasaka Y, Kakeya H, Fujita M, Hasegawa K, Morimoto T. Innovative preparation of curcumin for improved oral bioavailability. Biol Pharm Bull. 2011;34(5):660-5. doi: 10.1248/bpb.34.660. PMID 21532153
- [Result] Zaman MS, Chauhan N, Yallapu MM, Gara RK, Maher DM, Kumari S, Sikander M, Khan S, Zafar N, Jaggi M, Chauhan SC. Curcumin Nanoformulation for Cervical Cancer Treatment. Sci Rep. 2016 Feb 3;6:20051. doi: 10.1038/srep20051. PMID 26837852
- [Result] Dhillon N, Aggarwal BB, Newman RA, Wolff RA, Kunnumakkara AB, Abbruzzese JL, Ng CS, Badmaev V, Kurzrock R. Phase II trial of curcumin in patients with advanced pancreatic cancer. Clin Cancer Res. 2008 Jul 15;14(14):4491-9. doi: 10.1158/1078-0432.CCR-08-0024. PMID 18628464